CLINICAL TRIAL: NCT06174818
Title: Pulsed Radiofrequency Treatment Of the Gasserian Ganglion for tRigeminal nEuralgia: a retroSpective Study
Acronym: Progress
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Koen Van Boxem, principal investigator (MD PhD), Ziekenhuis Oost-Limburg
Other Study IDs: Z-2021102
Record Dates: First submitted 2023-09-07; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Trigeminal Neuralgia (TN)
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TN: Patients with trigeminal neuralgia
  Interventions: Procedure: PRF

INTERVENTIONS:
Procedure: PRF — Pulsed Radiofrequency Current of the Gasserian Ganglion

SUMMARY:
With the Pulsed Radiofrequency treatment (PRF) Of the Gasserian ganglion for tRigeminal nEuralgia: a retroSpective Study (PROGRESS) the objective is to document the outcome of PRF (Pulsed Radiofrequency treatment) for patients with TN (Trigeminal Neuralgia), unresponsive to conservative treatment.

DETAILED DESCRIPTION:
Primary objective:

To determine the proportion of patients in which PRF (pulsed radiofrequency) of the Gasserian ganglion for trigeminal neuralgia (TN) provides acute pain relief of at least 50% on the GPE (Global perceived effect) score (six weeks after treatment)

Secondary objectives:

- To determine the duration during which PRF of the Gasserian ganglion for trigeminal neuralgia provides a reduction of at least 50% on the GPE (Grade Point Equivalent) score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trigeminal neuralgia who underwent their first PRF of the Gasserian ganglion between 01/09/2013 and 31/08/2021

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with trigeminal neuralgia who underwent their first PRF of the Gasserian ganglion between 01/09/2013 and 31/08/2021
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
GPE <50% | Six weeks after treatment
  To determine the proportion of patients in which PRF (pulsed radiofrequency) of the Gasserian ganglion for trigeminal neuralgia (TN) provides acute pain relief of at least 50% on the GPE (Global perceived effect) score (six weeks after treatment)

SECONDARY OUTCOMES:
Duration of GPE <50% | From six weeks post procedure until definitive or possible relapse of neuralgia, assessed up to 48 months.
  To determine the duration during which PRF of the Gasserian ganglion for trigeminal neuralgia provides a reduction of at least 50% on the GPE (Grade Point Equivalent) score. This will be assessed six weeks post procedure and will be followed-up until definitive or possible relapse of neuralgia, assessed up to 48 months.

CONTACTS AND LOCATIONS:
Locations (1):
- ZOL Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium